CLINICAL TRIAL: NCT01796678
Title: Arginine Therapy in Sickle Cell Disease-VOC Clinical Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: HL 14386-05
Record Dates: First submitted 2013-02-19; First posted 2013-02-22 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Vaso-occlusive Pain Episodes
Keywords: sickle cell disease; vaso-occlusive pain episodes; arginine; nitric oxide
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Arginine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arginine (Experimental): 100 mg/kg T.I.D 3x a day IV or PO
  Interventions: Drug: Arginine
- Placebo (Placebo Comparator): Saline or sugar pill
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Arginine
  Other Names: L-arginine, L-arginine-HCL
  Arms: Arginine
Drug: Placebo — Saline or Sugar pill was given as placebo
  Arms: Placebo

SUMMARY:
Vaso-occlusion contributes significantly to morbidity in sickle cell disease (SCD). Vaso-occlusive painful episodes (VOE) are common and debilitating, causing the majority of emergency department visits. Currently efforts to treat painful episodes with use of non-steroidal pain relievers and intravenous narcotics offer symptomatic relief only, without targeting the underlying mechanisms of vaso-occlusion.Investigators have found that an arginine deficiency and low NO bioavailability occurs during painful events in SCD. Since arginine is the obligate substrate for NO production, and an acute deficiency is associated with VOE, investigators hypothesized that arginine supplementation may be a safe and beneficial treatment for sickle cell pain.

ELIGIBILITY:
Inclusion Criteria:

* Established Diagnosis of Sickle Cell Disease(SS,SC,S-beta thal)
* Admitted to Hospital for pain
* Pain requiring hospitalization for parenteral narcotics, not attributable to non-sickle cell causes
* >3 year and older

Exclusion Criteria:

* Hemoglobin less than 5gm/dL or immediate need for red cell transfusion
* Hepatic Dysfunction: increased in SGPT to >2x normal value
* Renal Dysfunction: increased in creatinine to >2x normal value or >1.5
* Mental status or neurological changes
* Pregnancy
* >10 Hospitalizations per year or history of dependance to narcotics
* Inability to take oral medications or allergy to arginine
* Inability to use a PCA device
* < 3 years of age

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2000-09; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Length of Hospital Stay | participants will be followed for the duration of hospital stay an expected average of 3-6 days, with re-admission data being collect for up to 30 days

SECONDARY OUTCOMES:
Effect on Pain Score | participants will be followed for the duration of hospital stay an expected average of 3-6 days
Total Opioid Use (mg/kg) | participants will be followed for the duration of hospital stay an expected average of 3-6 days

CONTACTS AND LOCATIONS:
Overall Officials: Claudia R Morris, MD, Principal Investigator — Childrens Hospital Oakland
Locations (1):
- Childrens Hospital Research Center Oakland, Oakland, California, United States

REFERENCES:
- [Result] Morris CR, Kuypers FA, Lavrisha L, Ansari M, Sweeters N, Stewart M, Gildengorin G, Neumayr L, Vichinsky EP. A randomized, placebo-controlled trial of arginine therapy for the treatment of children with sickle cell disease hospitalized with vaso-occlusive pain episodes. Haematologica. 2013 Sep;98(9):1375-82. doi: 10.3324/haematol.2013.086637. Epub 2013 May 3. PMID 23645695